CLINICAL TRIAL: NCT03778645
Title: Adrenal Venous Sampling Via an Antecubital Approach: A Multicenter Study
Brief Title: Adrenal Venous Sampling Via an Antecubital Approach
Acronym: AVSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2018-995
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Hyperaldosteronism; Angiography
Keywords: Adrenal venous sampling; Hyperaldosteronism; Angiography; Antecubital approach
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Adrenal Venous Sampling — Adrenal Venous Sampling via an Antecubital Approach

SUMMARY:
Currently, adrenal venous sampling (AVS) serves as the gold standard for subtyping of PA. Right adrenal vein catheterization is often difficult due to unfavorable anatomy of the vein including small vein size, short length, caudal direction for the transfemoral approach, and rare drainage to the accessory hepatic vein. All of these factors limit the widespread use of this approach. Given that the right adrenal vein is angled caudally in most patients, AVS via an antecubital approach was performed since January 2012. The purpose of this multicenter retrospective study was to evaluate the safety and feasibility of AVS via the antecubital approach.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is recognized as the most common cause of secondary hypertension, with a prevalence of approximately 10% among unselected hypertensive populations. Subtype diagnosis is crucial because unilateral primary aldosteronism can be treated by laparoscopic adrenalectomy or open surgery, which may result in a cure or significant improvement of blood pressure, thus decreases the incidence of cardio-cerebrovascular complications. Currently, adrenal venous sampling (AVS) serves as the gold standard for subtyping of PA. Given that the right adrenal vein is angled caudally in most patients, AVS via an antecubital approach was performed since January 2012 at the Fuwai Hospital. So far, there have been more than fifteen hospitals to have some experience on AVS via antecubital approach with investigators' helps. The purpose of this multicenter retrospective study was to evaluate the safety and feasibility of AVS via the antecubital approach.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the principal investigator to participate to the data collection of patients with primary aldosteronism underwent AVS via antecubital approach

Exclusion Criteria:

* Refusal of the principal investigator to participate to the AVSA Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with primary aldosteronism underwent AVS via antecubital approach between January 1st 2012 and December 31st 2018 in medical centers (agreement of the principal investigator to participate to the AVSA) in China
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of bilateral adrenal sampling | From January 1st 2012 to December 31st 2018

SECONDARY OUTCOMES:
The success rate of right adrenal sampling | From January 1st 2012 to December 31st 2018
The success rate of left adrenal sampling | From January 1st 2012 to December 31st 2018
The incidence of adrenal vein ruptures occurring during AVS | From January 1st 2012 to December 31st 2018

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease
Locations (10):
- China (10):
  - Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Eighth Affiliated Hospital of Sun Yat-sen University, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xi'an NO.3 Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Medical College of Shihezi Universtiy, Shihezi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong H, Huang J, Zhang Y, Dong Y, Liu M, Yan Z, Li J, Chen Y, Zou Y, Wang J, Kang Y, Jiang Z, Song W, Zuo Y, Xiong H, Xu J, Jiang X. Adrenal Venous Sampling Via an Antecubital Approach in Primary Aldosteronism: A Multicenter Study. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e274-e279. doi: 10.1210/clinem/dgad433. PMID 37466201